CLINICAL TRIAL: NCT06775275
Title: A Randomized Phase II Study of Adebrelimab in Combination with Chemotherapy with or Without Bevacizumab Neoadjuvant Therapy for Resectable Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Adebrelimab in Combination with Chemo with or Without Bevacizumab Neoadjuvant Therapy for Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Director, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-II
Record Dates: First submitted 2024-11-18; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Resectable Lung Non-Small Cell Carcinoma
MeSH Terms: interventions — Bevacizumab; Platinum Compounds; Paclitaxel; Docetaxel; Pemetrexed; Carboplatin; Cisplatin; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- four-drug combination group (Experimental): PD-L1 inhibitor with chemotherapy with Antiangiogenic therapy for neoadjuvant therapy
  Interventions: Drug: Adebellizumab; Drug: Bevacizumab; Drug: Platinum-based chemotherapy
- three-drug combination group (Experimental): PD-L1 inhibitor with chemotherapy for neoadjuvant therapy
  Interventions: Drug: Adebellizumab; Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: Adebellizumab — adebrelimab
Drug: Bevacizumab — bevacizumab
  Arms: four-drug combination group
Drug: Platinum-based chemotherapy — paclitaxel or albuminotaxol or docetaxel combined with platinum, pemetrexed combined with platinum. Platinums include carboplatin, cisplatin and nedaplatin.
  Other Names: paclitaxel; albuminotaxol; docetaxel; pemetrexed; carboplatin; cisplatin; nedaplatin

SUMMARY:
This is a prospective, multicenter, randomized, uncontrolled Phase II study to assess the efficacy and safety of adebrelimab in combination with chemotherapy with or without bevacizumab for the treatment of resectable Stage II-IIIB (T3N2) NSQ-NSCLC and to explore biomarkers associated with efficacy.

DETAILED DESCRIPTION:
Neoadjuvant therapy with experimental treatment followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Resectable NSQ NSCLC
* Age 18-65 years
* male or female
* ECOG 0-1
* Subjects have not received surgery, chemotherapy, radiotherapy and biological treatment of treatment-naive non-squamous non-small cell lung cancer
* Subjects must have adequate pulmonary function for the intended pneumonectomy;

Exclusion Criteria:

* SCLC or SQ NSCLC
* previously used anti-PD1, anti-PDL1, anti-CTLA4 antibodies, etc.
* patients who have previously used anti-angiogenic drugs;
* allergic to any component of the study drug or chemotherapy drugs
* patients with any severe and or uncontrolled disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | After 4 cycles of neoadjuvant therapy(3 weeks per cycle), surgical resection was performed at intervals of 4-6 weeks. Pathological response assessment results were assessed within one week after surgery.
  Pathological complete response, pCR (primary tumor + lymph nodes).It refers to the proportion of subjects with no residual surviving tumor cells (including lymph nodes) in the postoperative specimen among the enrolled subjects

SECONDARY OUTCOMES:
Major Pathological response | After 4 cycles of neoadjuvant therapy(3 weeks per cycle), surgical resection was performed at intervals of 4-6 weeks. Pathological response assessment results were assessed within one week after surgery.
  It refers to the proportion of subjects with residual surviving tumor cells of ≤ 10% in the postoperative specimen among the enrolled subjects.
Overall response rate | After 4 cycles of neoadjuvant therapy(3 weeks per cycle), before surgical resection was performed（at intervals of 4-6 weeks）.
  It refers to the proportion of patients whose tumor shrinks to a certain extent and maintains it for a certain period of time, including CR and PR cases.
event free survival | from randomization to imaging confirmation, local progression leading to inoperable tumors, unresectable tumors, local or distant recurrence, and death from any cause, whichever came first, assessed up to 24 months.
  Defined as disease progression from randomization to imaging confirmation, local progression leading to inoperable tumors, unresectable tumors, local or distant recurrence, and death from any cause.
safety | Safety follow-up will be conducted 30 ± 7 days after the last use of bevacizumab/chemotherapy or 90 ± 7 days after the last use of adebrelimab/surgery (whichever occurs later) to track the relief of AE. Incidence of AE/SAE/TRAE will be recorded.
  Monitoring and recording of adverse events, including Incidence of serious adverse events and adverse events of special interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No